CLINICAL TRIAL: NCT03917342
Title: Electroencephalographic Effects of Spinal Anaesthesia During Caesarean Delivery in Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: National Council of Scientific and Technical Research, Argentina (Other Government); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20190123
Record Dates: First submitted 2019-01-28; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Pre-Eclampsia; Effects of; Anesthesia, Spinal and Epidural, in Pregnancy
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Three groups of subjects studied: A: Control group: 15 healthy women B: 15 Healthy parturients: elective cesarean delivery C: 15 preeclamptic parturients: cesarean delivery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): EEG measure in 15 healthy women undergoing elective hysteroscopy under single shot spinal anesthesia. Bupivacaine 10mg (+-2mg) spinal dose with 15 mcg Fentanyl spinal dose
  Interventions: Device: EEG measure
- Healthy parturients (Active Comparator): EEG measure in 15 healthy parturients undergoing elective cesarean delivery under single shot spinal anesthesia.Bupivacaine 10mg (+-2mg) spinal dose with 15 mcg Fentanyl spinal dose
  Interventions: Device: EEG measure
- Preeclamptic parturients (Active Comparator): EEG measure in 15 parturients with preeclampsia undergoing elective cesarean delivery under single shot spinal anesthesia.Bupivacaine 10mg (+-2mg) spinal dose with 15 mcg Fentanyl spinal dose
  Interventions: Device: EEG measure

INTERVENTIONS:
Device: EEG measure — Frontal 3-derivation EEG measure under different conditions in pregnancy (healthy vs preeclampsia) and baseline non-pregnant women

SUMMARY:
Neuraxial anesthesia has been associated with delayed brainstem conduction and decreasing afferent sensory transmission, thereby modifying reticulo-thalamo-cortical mechanisms regulating arousal. The state of entropy measured by EEG-monitors has detected sedative effects associated with neuraxial anaesthesia in healthy volunteers, as well as during caesarean delivery. Entropy is a measure of the irregularity or disorder of a brains activity - sedation leading to a decrease of irregularity or disorder in the EEG.The aim of this pilot study is to prospectively assess the effect of spinal anaesthesia in healthy and preeclamptic parturients on brain activity. Decreased epileptiform activity in patients with preeclampsia would suggest that early neuraxial analgesia in labouring preeclamptic patients is beneficial, and may protect against neurological complications.

DETAILED DESCRIPTION:
Neuraxial anesthesia has been associated with delayed brainstem conduction and decreasing afferent sensory transmission, thereby modifying reticulo-thalamo-cortical mechanisms regulating arousal. The state of entropy measured by EEG-monitors has detected sedative effects associated with neuraxial anaesthesia in healthy volunteers, as well as during caesarean delivery. Entropy is a measure of the irregularity or disorder of a brains activity - sedation leading to a decrease of irregularity or disorder in the EEG.

The EEG activity in general can be separated into background activity, focal abnormalities, and intermittent and paroxysmal activity.8 Background electrical activity measured with the EEG by surface electrodes, are characterized by their corresponding frequency wave bands, ranging from slow waves (< 1 Hz), Delta (1 - 4 Hz), Theta (4 - 8 Hz), Alpha (8 - 12 Hz), Beta (12 - 30 Hz) and Gamma (> 30 Hz). In healthy volunteers, neuraxial anaesthesia was linked to increased activity - the so-called state of paradoxical excitation. This pattern is similar to the sedative low-dose GABAergic effects known to occur in response to the benzodiazepine midazolam. Epileptic potentials as paroxysmal EEG activity are typically seen with seizures, but they can be a sign of other changes of brain state as well (e.g. (pre)eclampsia or high doses of opioids).

Preeclampsia constitutes a heterogeneous multisystemic disorder defined by the new onset of hypertension and proteinuria after 20 weeks of gestation, affecting 2-8 % of all pregnancies world-wide. In this condition the nervous system is commonly affected, being the cause of significant morbidity and mortality, when seizures occur resembling an epileptic grand-mal convulsion. Significantly, cerebral white matter lesions are described several years after eclamptic episodes. Posterior reversible encephalopathy syndrome (PRES) is also suggested to be a core component of eclampsia. In this condition is associated extensive white matter changes have been detected, using advanced neuroimaging techniques. EEG changes can be detected before clinical signs of PRES are present, and before ischemia leads to irreversible brain damage.14 In preeclampsia EEG changes are also common, consisting of slow waves in the occipital lobe, as well as spike discharges. These EEG changes have been reported in eclampsia and in severe preeclampsia, with some differences between the two conditions. The prevention of eclampsia, which can occur pre-, intra-, or postpartum, is thus a critical management goal. Current literature only describes the use of EEG entropy - reflecting the state of arousal - during neuraxial anaesthesia in parturients. So far no study has assessed the quantitative (qEEG) or paroxysmal EEG changes induced by neuraxial anaesthesia in parturients undergoing caesarean delivery, and such monitoring has particular relevance in a high-risk patient population with preeclampsia.

Aims

The aim of this pilot study is to prospectively assess the effect of spinal anaesthesia in healthy and preeclamptic parturients on brain activity. Decreased epileptiform activity in patients with preeclampsia would suggest that early neuraxial analgesia in labouring preeclamptic patients is beneficial, and may protect against neurological complications.

ELIGIBILITY:
Inclusion Criteria:

* Group A: Healthy controls, American Society of Anesthesiology (ASA) I or II status, undergoing a hysteroscopic procedure under single shot spinal anaesthesia without intravenous or oral sedation.
* Group B:

  * Healthy ASA I or II status patients undergoing elective caesarean section at term (>37 weeks of gestation) under spinal single shot anaesthesia without intravenous or oral sedation.
  * Singleton pregnancy.
* Group C:

  * ASA I, II or III status patients undergoing elective secondary caesarean section at term (>37 weeks of gestation) under spinal single shot anaesthesia without intravenous or oral sedation
  * Singleton pregnancy
* Diagnosis of preeclampsia: Systolic blood pressure over140 mmHg or diastolic pressure over 90 mmHg and
* Proteinuria over 0.3 grams in a 24-hour urine or protein: creatinine ratio superior to 0.3 or signs of end-organ dysfunction (platelet count < 100,000 µL, serum creatinine >110 mg/L, or doubling of the serum creatinine, elevated serum transaminases to twice normal concentration)

Exclusion Criteria:

* Patient refusal.
* Active labour.
* Eclampsia.
* Hypertensive crisis as defined by systolic blood pressure over 210 mmHg or diastolic pressure over 120 mmHg.
* Known epilepsy.
* Anti-epileptic medication and magnesium sulphate.
* Reported or admitted medication or substance abuse (street drugs, opiates, benzodiazepines, alcohol).
* Known neurological condition with previously pathologic diagnostic imaging or EEG.
* Severe fetal malformations (gastroschisis and omphalocele, tracheo-oesophageal fistula, cerebral malformations in the category of cephalic disorders, pulmonary hypoplasia, congenital heart disease).
* Established rupture of membranes prior to spinal anaesthesia.
* Non-German and non-French speaking parturient.
* Lack of written consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender identity
Enrollment: 45 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Spectral analysis through fast Fourier transformation | Baseline, one minute and 60 minutes, 5 minutes for each measure
  Change from baseline EEG, EEG after one and 60 minutes after neuraxial anaesthesia
Spectral analysis of the detection of seizure activity by absolute slope analysis (composite endpoint) | Baseline, one minute and 60 minutes, 5 minutes for each measure
  Change from baseline EEG, EEG after one and 60 minutes after neuraxial anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Kaiser, MD, Study Chair — Bern University Hospital
Locations (1):
- Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No